CLINICAL TRIAL: NCT02483936
Title: Efficacy and Safety Evaluation of the New Association on Fixed Dose of Olmesartan Medoxomil + Chlorthalidone (40mg + 12.5mg and 40mg + 25mg) Compared With BENICAR HCT® in Hypertension Control
Brief Title: Efficacy and Safety of Olmesartan Associated With Chlorthalidone Versus Benicar HCT® in Essential Hypertension Control
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Decided by Sponsor
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OLCEMS0215
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension | interventions — Olmesartan Medoxomil; Chlorthalidone; olmesartan; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test 1: Olmesartan+Chlorthalidone (Experimental): The patients will take 1 tablet (Olmesartan medoxomil 40 mg + Chlorthalidone 12,5 mg) a day, in the morning.
  Interventions: Drug: Olmesartan medoxomil 40mg + chlorthalidone 12,5mg
- Test 2: Olmesartan+Chlorthalidone (Experimental): The patients will take 1 tablet (Olmesartan medoxomil 40 mg + Chlorthalidone 25 mg) a day, in the morning.
  Interventions: Drug: Olmesartan medoxomil 40mg + chlorthalidone 25mg
- Comparator 1: Benicar HCT® (Active Comparator): The patients will take 1 tablet (Olmesartan 40mg + Hydrochlorothiazide 12,5 mg) a day, in the morning.
  Interventions: Drug: Olmesartan 40mg + Hydrochlorothiazide 12,5mg
- Comparator 2: Benicar HCT® (Active Comparator): The patients will take 1 tablet (Olmesartan 40mg + Hydrochlorothiazide 25 mg) a day, in the morning.
  Interventions: Drug: Olmesartan 40mg + Hydrochlorothiazide 25mg

INTERVENTIONS:
Drug: Olmesartan medoxomil 40mg + chlorthalidone 12,5mg — 1 tablet a day
  Arms: Test 1: Olmesartan+Chlorthalidone
Drug: Olmesartan medoxomil 40mg + chlorthalidone 25mg — 1 tablet a day
  Arms: Test 2: Olmesartan+Chlorthalidone
Drug: Olmesartan 40mg + Hydrochlorothiazide 12,5mg — 1 tablet a day
  Other Names: Benicar HCT
  Arms: Comparator 1: Benicar HCT®
Drug: Olmesartan 40mg + Hydrochlorothiazide 25mg — 1 tablet a day
  Other Names: Benicar HCT
  Arms: Comparator 2: Benicar HCT®

SUMMARY:
The purpose of this study is to evaluate the non-inferiority clinical efficacy of two different drug associations in the essential hypertension control.

ELIGIBILITY:
Inclusion Criteria:

* Signed Consent of the patient;
* Participants with decompensated essential hypertension, classified into stage 1 (with high or very high cardiovascular risk), stage 2 or stage 3 according to the Brazilian Society of Cardiology (2010), who are being treated with monotherapy.

Exclusion Criteria:

* Patients with any clinically significant disease that in the investigator opinion can not participate in the study;
* Secondary hypertension diagnosis or blood pressure above 190x100 mmHg in the screening/randomization visit;
* Morbid obesity or immunocompromised patients;
* Participants with greater than 10 mmHg difference in the measurements of systolic or diastolic blood pressure between the two arms;
* Participants who do not have the two upper limbs;
* Participants with important electrocardiographic changes;
* Creatinine clearance - less than 60 mL / min;
* History of hypertensive emergencies and cardiovascular and / or moderate to severe cerebrovascular events in the past 6 months;
* Microalbuminuria urine sample greater than 30 mg/g;
* Patients with history of hypersensitivity to any of the formula compounds;
* Pregnancy or risk of pregnancy and lactation patients;
* Participation in clinical trial in the year prior to this study;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of essential hypertension control based on the reduction of systolic blood pressure at the end of the study. | 60 days

SECONDARY OUTCOMES:
Safety will be evaluated by the adverse events occurrences | 9 weeks
  Adverse events will be collected and followed in order to evaluate safety and tolerability